CLINICAL TRIAL: NCT05951296
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Investigate the Efficacy and Safety of Leramistat in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: A Study to Investigate Leramistat in Patients With IPF
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow initial recruitment and a lack of confidence in our ability to complete recruitment within the forecasted timeframe.
Sponsor: Modern Biosciences Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IST-07; 2023-504418-30 (EudraCT Number)
Record Dates: First submitted 2023-06-22; First posted 2023-07-19 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: IPF
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Leramistat (Experimental): Leramistat once daily
  Interventions: Drug: Leramistat
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Leramistat — Drug: Leramistat
  Arms: Leramistat
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
To compare the effect of daily oral dosing of leramistat over 12 weeks with placebo in participants aged 40 years or older with idiopathic pulmonary fibrosis (IPF).

DETAILED DESCRIPTION:
This will be a Phase 2, double-blind, placebo-controlled, 2-arm, parallel-group, multi-centre study to investigate leramistat treatment of patients aged 40 years or older with IPF. The study is planned to consist of the following parts:

Screening period: 1 to 28 days (Weeks -4 to -1). Treatment period: a 12-week blinded, placebo-controlled treatment period (Weeks 1 to 12).

Follow up period: 56 days (Weeks 13 to 20). All participants will return for a follow-up visit 56 days after their final dose.

Randomization will be stratified by concomitant use of an approved anti-fibrotic drug (nintedanib or pirfenidone) at randomization versus no concomitant use of an approved anti-fibrotic drug at randomization.

Number of Participants: Approximately 150 participants will be enrolled and randomly assigned in a 2:1 ratio to receive either leramistat or matched placebo.

If the participant is receiving nintedanib or pirfenidone treatment, it should be stable for at least 8 weeks prior to study entry and be predicted to remain stable during the course of the study. The maximum duration of participation (including screening period and follow-up) is 24 weeks.

Data Monitoring/Other Committee: A DSMB has been appointed for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of IPF based on: a. ATS/ERS/JRS/ALAT guidelines (Raghu, 2022) as confirmed by the investigator based on chest high-resolution computed tomography (hrCT) scan taken within 3 years of Screening and, if available, surgical lung biopsy b. UIP or probable UIP hrCT pattern consistent with the clinical diagnosis of IPF, as confirmed by central review prior to baseline (if indeterminate, hrCT findings of IPF may be confirmed locally by historical biopsy).
2. Has an FVC ≥45% of predicted.
3. Has a DLCO corrected for hemoglobin ≥25% and ≤80% of predicted.
4. Minimum distance on 6MWT of 150 meters.
5. Has a FEV1/FVC ratio >0.70.
6. If on anti-fibrotics, only the approved treatments of nintedanib or pirfenidone are allowed. Participants must be on a stable dose for at least 8 weeks prior to Visit 1
7. Has a life expectancy of at least 12 months (in the opinion of the investigator).

   * This list contains only key inclusion criteria.

Exclusion Criteria:

1. Emphysema ≥50% on hrCT or the extent of emphysema is greater than the extent of fibrosis according to the central reviewer's assessment from the most recent hrCT or if reported by the local reviewer.
2. Any current malignancy or a history of malignancy within the previous 5 years prior to screening, with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
3. Abnormality in heart rate, blood pressure or 12-lead ECG at screening that in the opinion of the Investigator increases the risk of participating in the study.
4. Significant history of drug allergy, including to leramistat or excipients, as determined by the Investigator.
5. Allergic reaction, anaphylaxis, or other reactions (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis or leukopenia)
6. History of opportunistic, chronic, or recurrent infections.
7. Participants with chronic obstructive pulmonary disease (COPD) or asthma that:

   * require >2 maintenance therapies
   * have experienced an exacerbation requiring hospitalization or systemic corticosteroids within 12 months prior to screening.

     * This list contains only key exclusion criteria.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Forced vital capacity (FVC) | 12 weeks
  Change from baseline in FVC versus placebo up to Week 12

OTHER OUTCOMES:
Adverse effects | 12 Weeks
  Incidence and frequency of treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Locations (56):
- United States (20):
  - UCSF Fresno, Fresno, California
  - National Jewish Health Main Campus, Denver, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Reliant Medical Research, Miami, Florida
  - US Associates in Research Inc, Miami, Florida
  - GCP Clinical Research, LLC, Tampa, Florida
  - GCP Clinical Research, Tampa, Florida
  - Southern Medical Research, LLC, Macon, Georgia
  - GenHarp Clinical Solutions, Chicago, Illinois
  - IU Health Ball Memorial Physicians Pulmonary and Critical Care Medicine, Muncie, Indiana
  - Benchmark Research - Covington - HyperCore - PPDS, Covington, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Howard County Center for Lung and Sleep Medicine, LLC, Columbia, Maryland
  - Hudson County Clinical Trials Research Center, Union City, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - Baylor Scott and White Health - Advanced Lung Disease Specialists - Dallas, Dallas, Texas
  - Metroplex Pulmonary and Sleep Medicine Center-4833 Medical Center Dr, McKinney, Texas
  - Metroplex Pulmonary and Sleep Medicine Centre 4833 Medical Center Dr, McKinney, Texas
  - University of Utah - PPDS, Salt Lake City, Utah
- France (4):
  - Hopital Nord AP-HM, Marseille
  - Hôpital Pasteur II, Nice
  - Hôpital Européen Georges Pompidou, Paris
  - Hopital Robert Schuman, Vantoux
- Germany (8):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Klinikum Köln-Merheim, Cologne
  - Ruhrlandklinik, Essen
  - IKF Pneumologie, Frankfurt am Main
  - Universitätsklinikum Gießen und Marburg GmbH, Giessen
  - Universitatsklinikum Halle (Saale), Halle
  - Universitatsklinikum Leipzig, Leipzig
  - Universitatsklinikum Schleswig-Holstein - Kiel, Lübeck
- Greece (7):
  - University Hospital of Alexandroupolis, Alexandroupoli
  - Evangelismos General Hospital of Athens, Athens
  - General Hospital of Diseases Thoracos of Athens "Sotiria", Athens
  - University General Hospital of Heraklion, Heraklion
  - University General Hospital of Ioannina, Ioannina
  - University General Hospital of Larissa, Larissa
  - Georgios Papanikolaou General Hospital of Thessaloniki, Thessaloniki
- Hungary (2):
  - Semmelweis Egyetem, Budapest
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- Israel (4):
  - Lady Davis Carmel Medical Center, Haifa
  - Rambam Medical Center - PPDS, Haifa
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center - PPDS, Tel Aviv
- Italy (5):
  - Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele, Catania
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Azienda Ospedaliero Universitaria Di Modena Policlinico, Modena
  - Fondazione Policlinico Universitario A Gemelli-Rome, Roma
  - Azienda Ospedaliera Universitaria Senese, Siena
- Spain (2):
  - Hospital Puerta del Mar, Cadiz
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (4):
  - Royal Brompton Hospital, London
  - University College Hospital, London
  - North Manchester General Hospital - PPDS, Manchester
  - Walsall Manor Hospital, Walsall